CLINICAL TRIAL: NCT03484221
Title: Totally Neoadjuvant FOLFOXIRI Chemotherapy Followed by Short-course Radiation and XELOX Chemotherapy in Patients With Locally Advanced Rectal Cancer：an Open-label, Single-arm, Multicenter Phase II Study.
Brief Title: Totally Neoadjuvant FOLFOXIRI + Short-course Radiation + XELOX in Patients With Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGIOG-2017-02
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Rectal Neoplasms; Drug Therapy; Radiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Fluorouracil; XELOX; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI+short-course radiation+XELOX (Experimental): Firstly, 4 cycles of neoadjuvant FOLFOXIRI chemotherapy were administered. Subsequently, a short-course radiation therapy (5Gy*5) will be performed. After that, 4 cycles of XELOX chemotherapy will be administered followed by surgery.
  Interventions: Drug: FOLFOXIRI; Radiation: Short-Course Radiation Therapy(5Gy*5); Drug: XELOX

INTERVENTIONS:
Drug: FOLFOXIRI — IRINOTECAN 150 mg/m^2 IV over 1-h, day 1 + OXALIPLATIN 85 mg/m^2 IV over 2-h, day 1 + L-LEUCOVORIN 200 mg/m^2 IV over 2-h, day 1 + 5-FLUOROURACIL 2800 mg/m^2 IV 48-h continuous infusion, starting on day 1 administered every two weeks for 4 cycles (2 months).
  Other Names: Irinotecan; Oxaliplatin; 5-Fluorouracil
Radiation: Short-Course Radiation Therapy(5Gy*5) — Patients received a short-course radiation therapy(5Gy*5) after 4 cycles of FOLFOXIRI.
Drug: XELOX — OXALIPLATIN 130 mg/m^2 IV over 2-h, day 1 Capecitabine 1000 mg/m^2 twice daily days 1-14 every 3 weeks for 4 cycles.
  Other Names: Capecitabine; Oxaliplatin

SUMMARY:
To evaluate the efficacy and safety of totally neoadjuvant FOLFOXIRI chemotherapy (irinotecan, oxaliplatin and fluorouracil) followed by short-course radiation therapy and XELOX chemotherapy in the patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiation therapy with double cytotoxic agents is the standard treatment for the patients with locally advanced rectal cancer. Conventional treatment reduced the local recurrence but did not prolong the long-term survival. Furthermore, the patients with pathological complete response (pCR) did not benefit from double cytotoxic chemotherapy. Therefore, we chose triple cytotoxic agents FOLFOXIRI as the neoadjuvant chemotherapy. We will evaluate the efficacy and safety of totally neoadjuvant FOLFOXIRI chemotherapy (irinotecan, oxaliplatin and fluorouracil) followed by short-course radiation and XELOX chemotherapy in the patients with locally advanced rectal cancer to achieve more pCR and longer survival.

In this prospective study, 30 patients with locally advanced rectal cancer will be recruited. Firstly, 4 cycles of neoadjuvant FOLFOXIRI chemotherapy were administered. Subsequently, a short-course radiation therapy (5Gy*5) will be performed. After that, 4 cycles of XELOX chemotherapy will be administered followed by TME surgery. PET-CT examination will be performed before and after the 4 cycles of neoadjuvant FOLFOXIRI chemotherapy to assess the SUVmax changes. In addition, the dynamic changes of ctDNA in peripheral blood will be monitored at the PET-CT examination. In the course of treatment, safety evaluation will be carried out according to the standard of adverse reaction classification (CTCAE) 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* Primary and pathological diagnosis of rectal adenocarcinoma
* Radiographic evaluation of initial resectable rectal cancer
* T staging was determined by MRI as T3N+ or T4Nx
* Distal border of the tumor must be located < 12 cm from the anal verge
* ECOG status: 0～1
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Neutrophil count≥1.5×10^9/L Platelet count≥90×10^9/L Hemoglobin≥90g/L Total bilirubin (TBI) ≤ 1.5 * ULN Alanine aminotransferase (ALT)≤2.5 * ULN Aspartate aminotransferase (AST)≤2.5 * ULN Alkaline phosphatase (ALP)≤2.5 * ULN

- Signed informed consent; able to comply with study and/or follow- up procedures

Exclusion Criteria:

* Previous treatment with oxaliplatin, irinotecan or fluorouracil
* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* Clear indication of involvement of the pelvic side walls by imaging
* With distant metastasis
* A history of malignant rectal cancer (i. e. sarcoma, lymphoma, carcinoid, squamous cell carcinoma) or synchronous colon cancer
* Cardiovascular disease that would preclude study treatment or follow-up; New York Heart Association class III or IV heart disease; active ischemic heart disease; myocardial infarction within the past 6 months; symptomatic arrhythmia uncontrolled hypertension. Unexplained syncope occurred within 3 months
* Digestive system diseases that would preclude study treatment or follow-up within the past 6 months
* Gastric ulcers or duodenal ulcers for the treatment of resistance;
* 3 or 4 grade gastrointestinal bleeding / bleeding;
* Gastrointestinal perforation / fistula;
* Abdominal abscess;
* Infectious or inflammatory bowel disease
* HIV infection and/or active hepatitis B virus infection
* Pregnant or lactating women. Fertile patients must use effective contraception
* Any serious acute or chronic disease that can not be involved in the study or to influence the interpretation of the results of the study
* Other intervention clinical trials were combined at the same time.
* Nerve or mental abnormality affecting cognitive ability
* Other malignancy except effectively treated squamous cell or basal cell skin cancer,
* Other situations that the researchers think should be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of tumor downstaging to stage 0 and stage I | 2 years
  Tumor downstaging from stage II or III to pathologic complete response (stage 0) and stage I

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | 2 years
  The level of tumor regression under pathological examination
Disease free survival | 3 years
  Estimated from the date of surgery to the date of recurrence.
Overall survival time | 3 years
  Estimated from the date of enrollment to death from any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 years
  The grade of toxicity will be assessed using the NCI-CTCAE version 4.0.
ctDNA change | 3 years
  The relationship between ctDNA and survival will be evaluated.
SUVmax changes | At the beginning of Cycle 1 and the end of Cycle 4 (each cycle is 14 days)
  Tumor metabolic response through FDG-PET examination before and after 4 cycles of neoadjuvant FOLFOXIRI chemotherapy
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 3 years
  Scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Jingdong Zhang, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Shenyang, China